CLINICAL TRIAL: NCT04272619
Title: LIVE-R Life: Liver Cancer Education
Brief Title: Liver Cancer Community Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-1039
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Liver Cancer
Keywords: prevention; education
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Cancer Education (Experimental)
  Interventions: Behavioral: LIVE-R Life Education

INTERVENTIONS:
Behavioral: LIVE-R Life Education — A health educator will present participants with a 30-minute PowerPoint presentation containing educational information about liver cancer risk, screening, prevention, symptoms, and treatments, as well as introduce the concept of neighborhood health (e.g., rates of liver cancer and related risk factors in a census tract and how that might influence individual cancer risk).

SUMMARY:
This study proposes to bridge the gap between evidence and action and combat rising liver cancer rates attributed to Hepatitis B and C infection in Philadelphia by identifying neighborhoods with higher than expected rates of liver cancer and related risk factors and administering an educational intervention about liver cancer and neighborhood health in those communities, working with existing community partners at Fox Chase Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Speaks/reads English
* Lives in Philadelphia or receives healthcare at a community partner site in Philadelphia

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liver Cancer Education
Started | 67
Completed | 67
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.25 (18.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 21
  More than one race | 2
  Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Liver Cancer Knowledge
Description: Liver cancer knowledge will be measured through four true/false items. Responses will be summed for a total liver cancer knowledge score. Score ranges run from 0-4, with higher scores indicating more knowledge. Change in knowledge is measured by subtracting baseline knowledge score from the post-intervention knowledge score. Change scores may range from -4 to 4, with positive scores indicating an increase in knowledge. Higher positive scores indicate a larger increase in knowledge.
Time Frame: Baseline, 30 minutes
Population: Five participants skipped the knowledge items on either the pre-test or the post-test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 62
score on a scale | 1.26 (1.09)

2. Primary Outcome: Change in General Interest in Learning About Neighborhood Health
Description: General interest in learning about neighborhood health will be measured through a single item asking, on a scale from strongly agree to strongly disagree, whether the participant would like to learn about liver cancer in their own neighborhood. Scores range from 1 to 5, with higher scores indicating more interest in learning about neighborhood health from a healthcare provider. Change in interest is measured by subtracting the baseline interest score from the post-intervention interest score. Change scores may range from -4 to 4, with positive scores indicating an increase in interest. Higher positive scores indicate a larger increase in interest.
Time Frame: Baseline, 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 67
score on a scale | -1.81 (1.50)

3. Primary Outcome: Change in Interest in Learning About Neighborhood Health From a Healthcare Provider
Description: Interest in learning about neighborhood health from a healthcare provider will be measured through a single item asking, on a scale from strongly agree to strongly disagree, whether the participant would like to learn about liver cancer in their own neighborhood from their doctor. Scores range from 1 to 5, with higher scores indicating more interest in learning about neighborhood health from a healthcare provider. Change in interest is measured by subtracting the baseline interest score from the post-intervention interest score. Change scores may range from -4 to 4, with positive scores indicating an increase in interest. Higher positive scores indicate a larger increase in interest.
Time Frame: Baseline, 30 minutes
Population: Two participants did not answer this item at pre- or post-test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 65
score on a scale | -0.95 (1.46)

4. Primary Outcome: Change in Interest in Learning About Neighborhood Health From Other Sources
Description: Interest in learning about neighborhood health from other sources will be measured through a single item asking, on a scale from strongly agree to strongly disagree, whether the participant would like to learn about liver cancer in their own neighborhood from non-medical sources (e.g., website or brochure). Scores range from 1 to 5, with higher scores indicating more interest in learning about neighborhood health from other sources. Change in interest is measured by subtracting the baseline interest score from the post-intervention interest score. Change scores may range from -4 to 4, with positive scores indicating an increase in interest. Higher positive scores indicate a larger increase in interest.
Time Frame: Baseline, 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 67
score on a scale | -0.90 (1.72)

5. Primary Outcome: Change in Interest in Discussing High Liver Cancer Risk With a Healthcare Provider
Description: Interest in discussing high liver cancer risk with a healthcare provider will be measured through a single item asking, on a scale from strongly agree to strongly disagree, whether the participant would be likely to discuss their liver cancer risk with a doctor if they learned they lived in a high-risk area. Scores range from 1 to 5, with higher scores indicating more interest in discussing liver cancer risk with a healthcare provider. Change in interest is measured by subtracting the baseline interest score from the post-intervention interest score. Change scores may range from -4 to 4, with positive scores indicating an increase in interest. Higher positive scores indicate a larger increase in interest.
Time Frame: Baseline, 30 minutes
Population: Three participants did not respond to this item at pre- or post-survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 64
score on a scale | -1.58 (1.69)

6. Primary Outcome: Change in Outcome Expectancies for Learning About Neighborhood Health - Patient Behavior
Description: Patient outcome expectancies for learning about neighborhood health will be measured through a single item asking, on a scale from 0 (not at all) to 10 (very much), whether learning about neighborhood health will help the participant make health decisions. Higher scores indicate more positive expectations. Change in outcomes expectancies is measured by subtracting the baseline score from the post-intervention score. Change scores may range from -10 to 10, with positive scores indicating an increase in outcome expectancies. Higher positive scores indicate a larger increase in expectations.
Time Frame: Baseline, 30 minutes
Population: One participant did not answer this item at pre- or post-survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 66
score on a scale | 0.83 (2.58)

7. Primary Outcome: Change in Outcome Expectancies for Learning About Neighborhood Health - Provider Behavior
Description: Provider outcome expectancies for learning about neighborhood health will be measured through a single item asking, on a scale from 0 (not at all) to 10 (very much), whether learning about neighborhood health will help the participant's healthcare provider make health decisions for them. Higher scores indicate more positive expectations. Change in outcome expectancies is measured by subtracting the baseline score from the post-intervention score. Change scores may range from -10 to 10, with positive scores indicating an increase in outcome expectancies. Higher positive scores indicate a larger increase in expectations.
Time Frame: Baseline, 30 minutes
Population: Two participants did not respond to this item at pre- or post-survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 65
score on a scale | -0.77 (2.40)

8. Primary Outcome: Change in Intentions About Communicating With Healthcare Provider - Neighborhood Prevalence of Liver Cancer
Description: intentions about communicating with healthcare provider about neighborhood liver cancer will be measured through a single item asking, on a scale from very likely to not at all likely, how likely the participant is to discuss liver cancer in their neighborhood with their healthcare provider over the next 12 months. Scores range from 1 to 5, with higher scores indicating higher likelihood of talking to a healthcare provider. Change in intentions is measured by subtracting the baseline score from the post-intervention score. Change scores may range from -4 to 4, with positive scores indicating an increase in intentions. Higher positive scores indicate a larger increase in intentions.
Time Frame: Baseline, 30 minutes
Population: One participants did not answer this item at pre- or post-survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 66
score on a scale | 0.79 (1.06)

9. Primary Outcome: Change in Intentions About Communicating With Healthcare Provider - Liver Cancer Screening
Description: intentions about communicating with healthcare provider about liver cancer screening will be measured through a single item asking, on a scale from very likely to not at all likely, how likely the participant is to discuss liver cancer screening with their healthcare provider over the next 12 months. Scores range from 1 to 5, with higher scores indicating higher likelihood of talking to a healthcare provider. Change in intentions is measured by subtracting the baseline score from the post-intervention score. Change scores may range from -4 to 4, with positive scores indicating an increase in intentions. Higher positive scores indicate a larger increase in intentions.
Time Frame: Baseline, 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 67
score on a scale | 0.67 (1.24)

10. Primary Outcome: Change in Intentions About Communicating With Healthcare Provider - Liver Cancer Risk
Description: intentions about communicating with healthcare provider about liver cancer risk will be measured through a single item asking, on a scale from very likely to not at all likely, how likely the participant is to discuss their personal risk factors for liver cancer with their healthcare provider over the next 12 months. Scores range from 1 to 5, with higher scores indicating higher likelihood of talking to a healthcare provider. Change in intentions is measured by subtracting the baseline score from the post-intervention score. Change scores may range from -4 to 4, with positive scores indicating an increase in intentions. Higher positive scores indicate a larger increase in intentions.
Time Frame: Baseline, 30 minutes
Population: Four participants did not respond to this item at pre- or post-survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liver Cancer Education
Number analyzed (Participants) | 63
score on a scale | 0.35 (0.97)

ADVERSE EVENTS:
Time Frame: One hour
Arm/Group | Liver Cancer Education
All-Cause Mortality (participants affected / at risk) | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT04272619/Prot_SAP_000.pdf